CLINICAL TRIAL: NCT04935723
Title: Cukurova University
Brief Title: The Effects of Reiki on Abdominal Surgery Patients' Anxiety, Fear, Postoperative Pain and Life Findings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Hamide Sisman, Principal Investigator., Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: G-5097-2020
Record Dates: First submitted 2021-06-10; First posted 2021-06-23 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Anxiety; Fear; Postoperative Pain; Reiki; Vital Signs
MeSH Terms: conditions — Anxiety Disorders; Pain, Postoperative | interventions — Therapeutic Touch

STUDY DESIGN:
Intervention Model Description: The study was planned as a three-group interventional randomized controlled study to examine the effect of Reiki touch therapy, which is a complementary method in relieving surgical fear, pain and anxiety in patients who will undergo open abdominal surgery.
Who Masked: Participant
Masking Description: The patients who will form the experimental group will not be told which method (reiki, sham reiki) will be applied.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EFFECT OF REIKIN ON ANXIETY, FEAR, PAIN AND LIFE FINDINGS OF ABDOMINAL SURGERY PATIENTS (Experimental): According to randomization, the patients in the reiki/sham reiki group were taken to a quiet single room and reiki/sham reiki was applied for approximately 25-30 minutes. will be applied. Reiki application will be applied by a researcher who has Reiki I and Reiki II level training.
  Interventions: Other: Reiki
- EFFECT OF SHAM REIKIN ON ANXIETY, FEAR, PAIN AND LIFE FINDINGS OF ABDOMINAL SURGERY PATIENTS (Placebo Comparator): According to randomization, the patients in the sham reiki group were taken to a quiet single room and sham reiki was applied for approximately 25-30 minutes. will be applied. Sham Reiki will be applied by a health professional who has not received Reiki training.
  Interventions: Other: Reiki
- ANXIETY, FEAR PAIN LEVELS AND LIFE FINDINGS OF ABDOMINAL SURGERY PATIENTS (No Intervention): The control group will be given routine post-operative care without any intervention and the data collection tools will be applied at the same time as the experimental group, twice at 30-minute intervals.

INTERVENTIONS:
Other: Reiki — The study was conducted as a three-group interventional randomized controlled trial to examine the effect of Reiki touch therapy on surgical fear, pain, anxiety and vital signs in patients undergoing open abdominal surgery. Reiki was applied to the first group and sham reiki to the second group. Group 3 formed the control group.
  Arms: EFFECT OF REIKIN ON ANXIETY, FEAR, PAIN AND LIFE FINDINGS OF ABDOMINAL SURGERY PATIENTS; EFFECT OF SHAM REIKIN ON ANXIETY, FEAR, PAIN AND LIFE FINDINGS OF ABDOMINAL SURGERY PATIENTS

SUMMARY:
Abdominal surgeries are those in which pain is felt severely due to the incision close to the diaphragm and an intensive neural network in the abdominal area. If the patient's post-operative pain is not controlled; Since it will restrict patient mobility, it can cause problems on many systems such as the pulmonary, cardiovascular and neuroendocrine system, and even suppress the immune system. Surgical intervention decision can cause anxiety in individuals regardless of the type of surgical procedure. Fear of anesthesia, fear of death, possibility of developing complications after surgery, pain, change in daily life activities, loss of social life and loss of control can lead to anxiety. In addition to all these, factors such as pain, fear, anxiety that stimulate the sympathetic nervous system can increase the pulse rate, blood pressure and respiratory rate.

Reiki, a complementary and alternative medicine (TAT) method, is a bioenergy based on the energy use of the body and has been used in various cultures for centuries in preventing and treating some diseases. Reiki is thought to help balance the body's natural energetic systems and reduce anxiety by transferring the available energy through hands. During Reiki, the activity of the parasympathetic system increases, pain and anxiety decrease. Thus, the patient's complaints are reduced by providing early discharge with possible complications after surgery.

Studies on the effectiveness of reiki, which is increasing worldwide use and recommended as a treatment approach for health services, are insufficient. The aim of this study, which is planned as a three-group interventional randomized control, is to examine the effect of reiki application on patients' negative reflections on pain, anxiety, fear and vital signs, which is the major surgery type in which patients experience the most pain.

DETAILED DESCRIPTION:
In line with the results of the power analysis using the Gpower 3.1.9.2 program, it was planned to include 31 patients in reiki, 31 patients in sham reiki and 31 patients in the control group, and the simple randomization method was used to distribute the sample to the study groups. Research data were collected in a quiet single room in the operating room Pre-op Unit and in the patient rooms of General Surgery I and II Clinics between July 2020 and December 2020. In order to determine the clarity of the data collection form, after obtaining permission from the ethics committee and pre-application with 12 patients who met the study criteria, "Personal Information Form", "Patient Follow-up Form" and Postoperative Period Patient Analgesic Follow-up Form" and "Reiki-Related Feedback Form" were prepared. filled. Application" Data were collected before and after reiki in the Pre-op unit on the 0th day before the operation, and in the General Surgery I and II clinics on the 1st and 2nd days after the operation. After obtaining the consent of the patient in the preoperative unit, the Personal Information Form, the Surgical Fear Scale and the STAI-I State Anxiety Scale were applied, and the results and vital findings after SPO2 were recorded in the Patient Follow-up. Form. According to randomization, the patients in the reiki/sham reiki group were taken to a quiet single room and reiki/sham reiki was applied for approximately 25-30 minutes. Done. Reiki application was applied by a researcher who received Reiki II level training, and sham reiki was applied by a health professional who did not receive reiki training. A written protocol is provided to both the Reiki practitioner and Sham Reiki practitioner describing hand positions, areas of practice, sequence and times. 5 minutes after the end of the application, the "Surgical Fear Scale" and the "STAI-I State Anxiety Scale" were re-administered, the patient's SPO2 and vital signs were taken again. In the control group according to randomization. The "Surgical Fear Scale" and the "STAI-I State Anxiety Scale" were applied and the patient's vital signs and SPO2 were measured. 30 minutes from assessment. Then, all measurements were repeated and recorded on the Patient Follow-up Form.

On the 1st and 2nd postoperative days, 4 hours after the routine analgesic drug administration, pulse, respiratory rate, blood pressure and SPO2 were measured and recorded in the patient follow-up form. After assessing the severity of pain with the "Visual Comparison Scale" and the anxiety with the "STAI-I State Anxiety Inventory", the patient was evaluated once a day for 25-30 minutes, depending on the group he was in. minute reiki/sham reiki was applied. 5 minutes after the end of the application. Then, the patient's pulse, respiratory rate, blood pressure and SPO2 were measured again and recorded in the Patient Follow-up Form. The severity of pain was re-evaluated with the "Visual Comparison Scale" and the state anxiety level with the "STAI-I State Anxiety Inventory". The analgesic doses/numbers used on the 1st and 2nd days were recorded in the "Analgesic Usage Follow-up Form". Routine postoperative care was given to the control group without any intervention, and data collection tools were applied at the same time as the experimental group twice at 30-minute intervals. After the final evaluation on the 2nd day, Reiki and Sham Reiki were applied to the group, and the "Reiki Application Feedback Form" was applied.

Statistical analyzes were performed using a package program called SPSS (IBM SPSS Statistics 24). Frequency tables and descriptive statistics were used to interpret the findings. Parametric methods were used for measurement values suitable for normal distribution. The "Independent Sample-t" test (t-table value) was used and the "ANOVA" test (F-table value) method was used to compare the measurement values of two independent groups in accordance with parametric methods. Compare the measurement values of three or more independent groups. The "Paired Sample-t" test (t-table value) method was used to compare the measurement values of the two dependent groups. Non-parametric methods were used for the measurement values that did not fit the normal distribution. "Mann-Whitney U" test (Z-table value) and "Kruskal-Wallis H" test (χ2-table value) were used to compare the measured values of two independent groups in accordance with non-parametric methods. ) method was used to compare the measurement values of three or more independent groups. . The "Wilcoxon" test (Z-table value) method was used to compare the measurement values of the two dependent groups.

ELIGIBILITY:
Inclusion Criteria:

No vision-hearing problems Able to communicate verbally No diagnosed psychologist problems Has past or present don't use of substances who will receive general anesthesia, ASA I, II and III, Elective open abdominal surgery,

Exclusion Criteria:

Patient Controlled Analgesia (PCA) use Those who have previously taken energy therapies such as Reiki Touch Therapy / Therapeutic Touch / Healing Touch who have had previous abdominal surgery,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-12-25 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 0-2 day
  Change of anxiety, fear, postoperative pain and vital signs of Reiki application before and after application.

CONTACTS AND LOCATIONS:
Overall Officials: Sevban Arslan, Phd, Study Chair — Çukurova University Faculty of Health Sciences Adana, Turkey
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The doctorate will be decided after the thesis defense